CLINICAL TRIAL: NCT01508351
Title: The Hypotensive Effect of Propofol: an Observational Study of Hypotension With Anesthetic Induction by Propofol in the General Population Under Standard of Care Anesthesia
Brief Title: The Hypotensive Effect of Propofol: an Observational Study
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Verbeek, Assistant Professor, Anesthesiology, Milton S. Hershey Medical Center
Other Study IDs: 38444
Record Dates: First submitted 2012-01-09; First posted 2012-01-11 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Hypotension; Anesthesia
Keywords: Propofol; Induction; Hypotension; General population
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Propofol Induction: All patients receiving propofol induction of anesthesia who are ASA 1-3

SUMMARY:
Hypotension is a recognized frequent complication of induction of anesthesia. The intent of this research is to determine the incidence of hypotension in patients receiving anesthetic induction with propofol. This investigation seeks to examine how normal clinical practice or a "real world" understanding of the usual response to propofol affects hemodynamics without isolating or standardizing other variables. The current research concerns hypotension in normal clinical practice where variability exists. This project aims to gather information and data in an attempt to form a foundation upon which each of the other variables affecting blood pressure may be subsequently assessed.

ELIGIBILITY:
Inclusion Criteria:

* All ASA 1-3 patients who are to receive propofol induction for general anesthesia

Exclusion Criteria:

* Allergy to propofol
* ASA 4 and above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hershey Medical Center patients presenting for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The systolic, diastolic, and mean arterial pressure. | Within first 20 minutes after anesthesia induction
  The systolic, diastolic, and mean arterial pressure will be measured every minute for twenty minutes. Blood pressure readings of Mean Arterial Pressure less than 65mmHg, Systolic Blood Pressure less than 80mmHg, or Diastolic Blood Pressure less than 40mmHg will be considered as hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States